CLINICAL TRIAL: NCT01963884
Title: Study of Tooth Alveolar Extraction Socket Anatomy and Its Relation to Alveolar Post-extraction Changes
Brief Title: Relate Tooth Alveolar Extraction Socket Anatomy to Alveolar Remodeling Rate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Implantology Institute (Other)
Responsible Party: Principal Investigator, Andre Chen, Msc, Implantology Institute
Other Study IDs: II-04
Record Dates: First submitted 2013-10-12; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Loss of Teeth Due to Extraction; Alveolar Bone Loss; Bone Resorption
Keywords: Extraction Sockets; Ridge dimensions; Dental Alveolar Anatomy; Dental Implants; Bone Physiology
MeSH Terms: conditions — Alveolar Bone Loss; Bone Resorption | interventions — Tooth Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Alveolar Socket Below Basal Bone: Tooth and the alveolar socket are positioned below basal bone. Measure Alveolar Socket remodeling, after Tooth Extraction with cone-beam technology evaluation
  Interventions: Procedure: Tooth Extraction; Radiation: Cone-Beam technology evaluation; Other: Measure Alveolar Socket Remodeling
- Alveolar Socket in Basal Bone (imbedded): Tooth and alveolar socket are positioned in basal bone. Measure Alveolar Socket remodeling, after Tooth Extraction with cone-beam technology evaluation
  Interventions: Procedure: Tooth Extraction; Radiation: Cone-Beam technology evaluation; Other: Measure Alveolar Socket Remodeling
- Alveolar Socket Buccal to Basal Bone: Tooth and alveolar socket are positioned buccally in relation to maxillary basal bone. Measure Alveolar Socket remodeling, after Tooth Extraction with cone-beam technology evaluation
  Interventions: Procedure: Tooth Extraction; Radiation: Cone-Beam technology evaluation; Other: Measure Alveolar Socket Remodeling

INTERVENTIONS:
Procedure: Tooth Extraction — Tooth from the maxillary anterior area extracted and alveolar socket remains intact
Radiation: Cone-Beam technology evaluation — Patient is submitted to a localized cone-beam image before tooth extraction and 6 month later, prior to implant installation.
  Other Names: Computerized Tomography; Imaging exams
Other: Measure Alveolar Socket Remodeling — In a computer, cone-beam images are superimposed to measure total the amount of ridge dimension
  Other Names: Digital Measurements

SUMMARY:
In patients that are going to be subjected to a tooth extraction in the anterior maxillary (from canine to canine) does the position of the intact alveolar socket related to maxillary basal bone interferes with the rate of resorption and remodeling process of the alveolar ridge ?

DETAILED DESCRIPTION:
We intend to demonstrate the physiologic process of the post-extraction socket and we hypothesized that the position of the socket in relation to basal bone, may project the remodeling process through three different equations.

A- tooth-periodontal apparatus is placed buccally of the basal bone - Equation 1

Anatomy Features- only 1-2 mm of lamina dura on the buccal part, 1-2mm of lamina dura on the palatal, plus basal bone.

Physiologic features - when the alveolar apparatus remodels, after tooth extraction, the amount that we project for resorption is : 1-2 mm of buccal lamina dura, the buccal-palatal dimension of the tooth that was extracted plus the 1-2 mm of palatal lamina dura.

At 6 month we hypothesized that 3 mm of trabecular bone may be present, so we may account for 2-3 mm more.

Due to conical anatomy of anterior teeth, the amount of trabecular bone will be more pronounced in the coronal area than in apical area, so we also account for that variation.

At this stage we project that the amount of ridge dimension will be :

buccal soft tissue (BST) + trabecular alveolar bone (ATB) + basal bone (BB) + palatal soft tissue (PST) Equation at 6 Month = (BST + ATB + PST).

But at 1 year the trabecular bone may be absent, so we project that the equation will be :

buccal soft tissue+basal bone+palatal soft tissue. Equation at 1 Year (BST + BB + PST)

at the end, ridge dimension will be : palatal basal bone plus soft tissue buccally and palatally.

Numbers for Buccal placed alveolus apparatus :

At Pre-extraction appointment (estimate) :

BST+ Lamina Dura Buccal + tooth buccal lingual dimension + palatal lamina dura + BB + PST (3mm + 1mm + X+ 1mm + Y + 3mm) = 8 mm + X (a or b or c) + Y (a or b or c)

X = For Anterior Teeth= 3 measures = coronal (Xa) + middle (Xb) + apical (Xc) Y- Basal bone is genetically predetermined and vary from person to person but geometrically can have two measures one middle (Ya) and one apical (Yb)

Note : the buccal-lingual dimensions vary from coronal to apical (either in the tooth root and in basal bone), so we hypothesize that the subtraction from pre-extraction values to post-extraction will more pronounced in coronal area than in the apical area.

At 6 month post-extraction :

BST+ ATB (varies coronal (a) , middle (b) , apical (c)) + BB + PST (3mm + ATB (a or b or c) + Y + 3mm) = 6 mm + ATB (a or b or c) + Y (a or b)

At 1 Year post-extraction

BST + BB + PST (3mm + X1 + 3mm) = 6 mm + Y (a or b )

Example For Central Incisor :

Before Extraction (estimate)

at coronal part pre-extraction : 3 + 1 + 10 (Xa) + 1 + 3 (Ya) + 3 = 21 mm at middle part pre-extraction : 3 + 1 + 5 (Xb) + 1 + 5 (Yb) + 3 = 18 mm at apical part pre-extraction : 3 + 1 + 2 (Xc) + 1 + 8 (Yc) + 3 = 18 mm

After Extraction 6 month (estimate)

at coronal part post-extraction : 3 + 3 (ATBa) + 3 + 3 = 12 mm at middle part post-extraction : 3 + 2 (ATBb) + 5 + 3 = 13 mm at apical part post-extraction : 3 + 1 (ATBc) + 8 + 3 = 15 mm

Variation expected (estimate) from Pre-extraction to 6 month post-extraction in buccally placed alveolar socket will be (estimate):

At coronal part ⨺ (variation) = 9 mm (43% reduction) at middle part ⨺ (variation) = 5 mm (28% reduction) at middle part ⨺ (variation) = 3 mm (17% reduction)

After Extraction 1 Year (estimate)

at coronal part post-extraction : 3 + 3 + 3 = 9 mm at middle part post-extraction : 3 + 5 + 3 = 11 mm at apical part post-extraction : 3 + 8 + 3 = 14 mm

Variation expected (estimate) from Pre-extraction to 1 year post extraction in buccally placed alveolar socket will be:

At coronal part ⨺ (variation) = 12 mm (57% reduction) at middle part ⨺ (variation) = 7 mm (39% reduction) at middle part ⨺ (variation) = 4 mm (22% reduction)

B- Tooth-periodontal apparatus is inferior of the basal bone (true socket) - Equation 2

Anatomy features- only 1-2 mm of lamina dura on the buccal and palatal part, no basal bone palatal, the basal bone is superior to the alveolar process.

Physiologic features - when the alveolar apparatus remodels after tooth extraction we project that the amount of resorption will be 1-2 mm of buccal lamina dura, the buccal-palatal dimension of the tooth that was extracted, plus the 1-2 mm of palatal lamina dura.

At 6 month, we hypothesized that 3 mm of trabecular bone may be present, so we may account for 2-3 mm more. At this stage the amount of ridge dimension will be composed by :

buccal soft tissue (BST) + trabecular alveolar bone (ATB) + palatal soft tissue (PST), (BST+ATB+PST).

note : lamina dura disappears, but because periosteum has to adhere to bone an outer cortical forms that surrounds remaining trabecular bone.

Numbers for Inferior placed alveolus apparatus :

At Pre-extraction appointment (estimate) :

BST+ Lamina Dura Buccal + tooth buccal-lingual dimension + palatal lamina dura + PST Equation = (3mm + 1mm + X+ 1mm + 3mm) = 8 mm + X (a or b or c)

X = For Anterior Teeth = 3 measures = coronal (Xa) + middle (Xb) + apical (Xc)

note : the buccal-lingual dimensions vary from coronal to apical (either in the tooth root and in basal bone), so we hypothesize that the subtraction from pre-extraction values to post-extraction will more pronounced in coronal area than in the apical area

At 6 month post-extraction (estimate) :

BST+ ATB (varies coronal (a) , middle (b) , apical (c) + PST Equation = (3mm + ATB (a or b or c) + 3mm) = 6 mm + ATB (a or b or c)

At 1 Year post-extraction (estimate)

BST + ATB (a or b or c) + PST (3mm + X1 + 3mm) = 6 mm + ATB (a or b or c)

Example For Central Incisor :

Before Extraction (estimate)

at coronal part pre-extraction : 3 + 1 + 10 (Xa) + 1 + 3 = 18 mm at middle part pre-extraction : 3 + 1 + 5 (Xb) + 1 + 3 = 13 mm at apical part pre-extraction : 3 + 1 + 2 (Xc) + 1 + 3 = 10 mm

After Extraction 6 month (estimate)

at coronal part post-extraction : 3 + 3 (ATBa) + 3 = 9 mm at middle part post-extraction : 3 + 2 (ATBb) + 3 = 8 mm at apical part post-extraction : 3 + 1 (ATBc) + 3 = 7 mm

Variation expected (projected) from Pre-extraction to 6 month post-extraction in inferior placed alveolar socket will be (estimate):

At coronal part ⨺ (variation) = 9 mm (43% reduction) at middle part ⨺ (variation) = 5 mm (28% reduction) at middle part ⨺ (variation) = 3 mm (17% reduction)

After Extraction 1 Year (estimate)

at coronal part post-extraction : 3 + 2 + 3 = 8 mm at middle part post-extraction : 3 + 2 + 3 = 8 mm at apical part post-extraction : 3 + 2 + 3 = 8 mm

Variation expected (estimate) from Pre-extraction to 1 year post-extraction in inferior placed alveolar socket will be:

at coronal part ⨺ (variation) = 10 mm (57% reduction) at middle part ⨺ (variation) = 5 mm (38% reduction) at middle part ⨺ (variation) = 2 mm (20% reduction)

C- tooth-periodontal apparatus is in (imbedded) the basal bone - Equation 3

Anatomy features- only 1-2 mm of lamina dura on the buccal part, 1-2mm of lamina dura on the palatal plus basal bone on the buccal and on the lingual part.

Physiologic features - when the alveolar apparatus remodels after tooth extraction, we project that the amount of resorption will be 1-2 mm of buccal lamina dura the buccal-palatal dimension of the tooth that was extracted plus the 1-2 mm of palatal lamina dura.

At 6 month, we hypothesized that 3 mm of trabecular bone may be present so we may account for 2-3mm more. At this stage the amount of ridge dimension will be composed by:

buccal soft tissue (BST) + Buccal basal bone (BBB) + trabecular alveolar bone (ATB)+ palatal basal bone (LBB)+ palatal soft tissue (PST), Equation = (BST+BBB+ATB+PBB+PST)

Numbers for Imbedded alveolus apparatus :

At Pre-extraction appointment (estimate):

BST+ BBB (Y1 a or b or c) + Lamina Dura Buccal + tooth buccal lingual dimension (X a or b or c) + palatal lamina dura + PBB (Y2 a or b or c or d) + PST (3mm + 1mm + X+ 1mm + 3mm) = 8 mm +Y1 + X (a or b or c or d) +Y2

X = For Anterior teeth = 3 measures = coronal (Xa) + middle (Xb) + apical (Xc)

Y1- Buccal Basal bone is genetically predetermined and vary from person to person geometrically 3 measures coronal (a) middle (b) and apical (c)

Y2- Palatal Basal bone (PBB) is genetically predetermined and vary from person to person geometrically 3 measures coronal (a) middle (b) and apical (c)

note : the buccal-lingual dimensions vary from coronal to apical (either in the tooth root and in basal bone), so we hypothesize that the subtraction from pre-extraction values to post-extraction will more pronounced in coronal area than in the apical area

At 6 month post-extraction (estimate):

BST+ BBB (Y1 a or b or c) + ATB (varies coronal (a) , middle (b) , apical (c)) + PBB (Y2 a or b or c) + PST (3mm + Y1+ ATB (a or b or c) + Y2 + 3mm) = 6 mm + ATB (a or b or c)

At 1 Year post-extraction (estimate)

BST+ BBB (Y1 a or b or c) + ATB (a or b or c) + PBB (Y2 a or b or c) + PST (3mm + X1 + 3mm) = 6 mm + Y1 (a or b or c) + ATB (a or b or c) + + PBB (Y2 a or b or c)

Example For Central Incisor :

Before Extraction (estimate)

at coronal part pre-extraction : 3 + 3 + 1 + 10 (Xa) + 1 + 3 + 3 = 24 mm at middle part pre-extraction : 3 + 5 + 1+ 5 (Xb) + 1 + 5 + 3 = 23 mm at apical part pre-extraction : 3 + 8 + 1 + 2 (Xc) + 1 + 8 + 3 = 26 mm

After Extraction 6 month (estimate)

at coronal part post-extraction : 3 + 3 + 10 (ATBa) + 3 + 3 = 22 mm at middle part post-extraction : 3 + 5 + 5 (ATBb) + 5 + 3 = 21 mm at apical part post-extraction : 3 + 8 + 2 (ATBc) + 8 + 3 = 24 mm

Variation expected (estimate) from Pre-extraction to 6 month post-extraction in imbedded placed alveolar socket will be:

At coronal part ⨺ (variation) = 2 mm (8% reduction) at middle part ⨺ (variation) = 2 mm (8% reduction) at middle part ⨺ (variation) = 2 mm (8% reduction)

After (estimate) Extraction 1 Year

at coronal part post-extraction : 3 + 3? + 10 + 3 ?+ 3 = 14 mm at middle part post-extraction : 3 + 5?+ 5 + 5? + 3 = 18 mm at apical part post-extraction : 3 + 8 ? + 2 + 8? + 3 = 8 mm

Variation expected (estimate) from Pre-extraction to 1 year post-extraction in imbedded placed alveolar socket will be:

At coronal part ⨺ (variation) = 2 mm (8% reduction) at middle part ⨺ (variation) = 2 mm (8% reduction) at middle part ⨺ (variation) = 2 mm (8% reduction)

ELIGIBILITY:
Inclusion Criteria:

* Patient that require a maxillary anterior extraction
* Sign Informed Consent
* Indication for a two-stage implant placement

Exclusion Criteria:

* Indication for immediate implants
* Indication for alveolar socket preservation or bone regeneration
* Indication for soft tissue graft
* Diabetes
* taking oral or intravenous biphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that require at least on tooth extraction of the upper anterior jaw (maxilla) canine, central incisor and lateral incisor.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Changes in alveolar ridge dimensions | From Tooth extraction (baseline T0) to T1 (6 month) to T2 (12 month)
  report the change in alveolar extraction socket dimensions from tooth extraction to 1 year, measured in digital computer, from Cone-Beam originated images.

CONTACTS AND LOCATIONS:
Overall Officials: Andre Chen, Msc, Principal Investigator — Implantology Institute; João Caramês, Phd, Study Director — Implantology Institute; Helena Francisco, Msc, Study Chair — Implantology Institute; Elena Cervino, Msc, Study Chair — Implantology Institute
Locations (1):
- Instituto de Implantologia, Lisbon, Lisbon District, Portugal